CLINICAL TRIAL: NCT05425498
Title: The Effects of Physical Activity Behavior Change in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hatice Nihan BOZKURT, Research Assistant, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6039-GOA
Record Dates: First submitted 2022-06-11; First posted 2022-06-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant Recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Program Group (Experimental): In the physical activity group, In the physical activity group, a 12-weeks physical activity program will be applied by giving pedometer. 12 telephone sessions will be held once a week according to motivational interview techniques based on the Transtheoretical Model. Assessments will perform just before starting to study, at the end of 12 weeks (just after the physical activity program), and the end of 24 weeks.
  Interventions: Other: Physical activity program
- Control group (No Intervention): In the control group, information about physical activity will be given without applying the physical activity program. Control group's assessments will be performed when they are included in the study, at the end of 12 weeks and 24 weeks.

INTERVENTIONS:
Other: Physical activity program — 12-weeks physical activity program will be applied by giving pedometer. 12 telephone sessions will be held once a week according to motivational interview techniques based on the Transtheoretical Model.
  Arms: Physical Activity Program Group

SUMMARY:
The aim of this study is to investigate the effects of physical activity program according to motivational interviewing based on the Transtheoretical Model on cardiovascular risk factors, physical activity level, physical activity behavior, and gait parameters in kidney transplant recipients.

DETAILED DESCRIPTION:
The Transtheoretical Model evaluates readiness for behavior change. The Transtheoretical Model has been frequently used to determine how individuals adopt and maintain physical activity. In kidney transplant recipients (KTRs), increased physical activity level is associated with better graft function, and decreased physical activity is associated with increased cardiovascular and all-cause mortality. Therefore, it is important to evaluate the level of physical activity and to gain physical activity habits in KTRs. The aim of this study is to investigate the effects of physical activity program according to motivational interviewing based on the Transtheoretical Model on on cardiovascular risk factors, physical activity level, physical activity behavior, and gait parameters in KTRs.

28 KTRs who meet the inclusion criteria will be assigned to the physical activity program or control group by non-randomization method. In the physical activity group, a 12-weeks physical activity program will be applied by giving pedometer. 12 telephone sessions will be held once a week according to motivational interview techniques based on the Transtheoretical Model. Assessments will perform just before starting to study, at the end of 12 weeks (just after the physical activity program), and the end of 24 weeks. In the control group, information about physical activity will be given without applying the physical activity program. Control group's assessments will be performed when they are included in the study, at the end of 12 weeks and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* to be at least 18 years old
* to have had a kidney transplantation at least 6 months ago

Exclusion Criteria:

* Pregnancy
* Multiple organ transplantation
* Severe cognitive impairment (Mini Mental Test score less than 24)
* Uncorrected visual impairment
* Certain neurological pathology (parkinson, stroke, epilepsy)
* Orthopedic surgery or injury to the lower extremity that will affect individuals' participation in daily life
* Inability to walk independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
HeartScore system | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  Assess cardiovascular risk.
Blood pressure | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  mmHg
Heart rate | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  beats per minute
Hemoglobin | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  g/dL
Body Mass Index | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  Body Mass Index is weight in kilograms divided by height in meters squared. Formula: weight (kg) / [height (m)]2
Lipid profile | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  total cholesterol level, LDL and HDL cholesterol, triglyceride (mg/dL)
Waist circumference | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  centimeter
C-reactive protein | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  mg/L
Glomerular filtration rate | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  ml/dk/1.73m2
Blood Glucose | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  mg/dL

SECONDARY OUTCOMES:
Physical activity monitor (SenseWear Armband) | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  Assess physical activity. Number of steps, total energy expenditure (calories), day and night average sleep time (minutes), day and night average lying time (minutes), average metabolic equivalent (MET), energy expenditure consumed during moderate-intensity (3 MET) physical activity (calories), physical activity time (minutes, 3 METs) results are obtained.
Exercise Stages of Change Questionnaire | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  Determines stages of physical activity behavior change. These stages of behaviour change consist of precontemplation, contemplation, preparation, action and maintenance.
G-Walk sensor system | Change from Baseline at 12 weeks, change from Baseline at 24 weeks, change from 12 weeks at 24 weeks
  Assess gait parameters. Gait parameters include gait speed (meters per second) and cadence (steps per minute).

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)